CLINICAL TRIAL: NCT05608096
Title: European Registry for Hemadsorption of Septic Patients With the Seraph 100 Microbind Affinity Blood Filter (ASTREA Study)
Brief Title: European Registry for Hemadsorption in Sepsis With the Seraph Filter
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Croatian Society for Organ Support (Other)
Collaborators: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Vedran Premuzic, Principal Investigator, Croatian Society for Organ Support
Other Study IDs: ASTREA-1982
Record Dates: First submitted 2022-10-26; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Sepsis; Acute Respiratory Distress Syndrome; Infections - Pathogen Unspecified; Disease; Critical Illness; Multi Organ Failure; Systemic Inflammatory Response Syndrome
Keywords: Acute Respiratory Distress Syndrome; Sepsis; Critical Illness; Multi Organ Failure; Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Sepsis; Respiratory Distress Syndrome; Disease; Critical Illness; Multiple Organ Failure; Systemic Inflammatory Response Syndrome | interventions — Hemoperfusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Hemoperfusion: ICU septic patients treated with hemoperfusion
  Interventions: Device: Hemoperfusion
- non-hemoperfusion: ICU septic patients non treated with hemoperfusion

INTERVENTIONS:
Device: Hemoperfusion — Commercial membrane for extracorporeal blood purification (hemoperfusion)
  Groups: Hemoperfusion

SUMMARY:
Although new techniques like extracorporeal blood purification have lately emerged, septic patients still have very high hospital mortality rates. Sepsis can be induced by either viremia, bacteriemia or in some cases both. Many studies have reported the effectiveness of different hemadsorbers, but patient sample sizes have been inadequate for definitive conclusions. Secondly, there are still no clear inclusion criteria as well as criteria for when to cease hemadsorption mostly due to immune dysregulation or cascade coagulation disorders. The aim of this observational prospective registry is to evaluate the effectiveness of the Seraph® 100 Microbind® Affinity Blood Filter (Seraph 100) in the treatment of septic ICU patients and to evaluate which cluster of these patients should benefit most with this therapy.

DETAILED DESCRIPTION:
Hemadsorption was introduced in everyday clinical practice before the COVID-19 pandemic. The efficacy of hemadsorption removal of endotoxins and cytokines is still, by some, controversial due to the fact that most of the studies were performed in a small number of patients with very different diagnoses, comorbidities and disease severity. Furthemore, some studies enrolled patients over a prolonged period of time with very high SOFA scores and multi-organ failure where it is difficult to expect any significant effect of any kind of organ support therapy. The COSA registry reported that the treatment of COVID-19 patients with Seraph 100 was well tolerated and observed lower mortality in the registry when compared to calculated mortality.

The primary aim of this observational prospective, multi-center, multistate web-based registry is to define the effectiveness and outcome of Seraph 100 treatment(s), investigate possible advantages of early targeted treatment and to set indications/inclusion criteria for the treatment of ICU septic patients with the method of hemoadsorption.

ELIGIBILITY:
Inclusion Criteria:

1. Sepsis or septic shock: sepsis is defined as the presence of suspected or documented infections along with systemic inflammatory response syndrome; septic shock is defined as the presence of sepsis and acute circulatory failure according to European criteria Society for Intensive Care Medicine
2. laboratory and clinical evidence of systemic inflammation: high levels of inflammatory cytokines such as IL-6 (>25 pg / ml); high values of inflammatory parameters from serum (leukocytes >15x10 9 / l, CRP >40 mg / l, procalcitonin >0.9 mg / l) and a high SOFA score (>2).
3. clinical symptoms of hemodynamic instability requiring vasopressors
4. diagnosis of ARDS
5. deterioration of respiratory status with the onset of respiratory failure requiring mechanical ventilation (respiration rate >30 / min, or oxygen saturation <93%, or PaO2 / FiO2 ratio <300mmHg).
6. Admission to ICU

Exclusion Criteria:

besides contraindications to the use of the hemoperfusion adopted (as from the manual of instructions), there are no exclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All medical institutions from European countries (Croatia, Finland, Germany, Italy, France, Greece, Slovenia) that provide extracorporeal blood purification treatments to septic critically ill patients are eligible for participation.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Survival | 28 days
  Overall Survival after Seraph 100 therapy session

SECONDARY OUTCOMES:
Define the inclusion criteria for hemoperfusion with Seraph 100 in ICU septic patients | 28 days
  Define the inclusion criteria for extracorporeal blood purification (hemoperfusion) with Seraph 100 in ICU septic patients
To assess the correlation between hemoperfusion and positive short-term outcome | Immediately after first hemoperfusion procedure
  Define as to assess the correlation between hemoperfusion and positive short-term outcome (i.e. an improvement in hemodynamic stability and respiratory status will be combined to report SOFA score)
To assess the correlation between hemoperfusion and positive short-term outcome | Immediately after first hemoperfusion procedure
  Define as to assess the correlation between hemoperfusion and positive short-term outcome (i.e. an improvement in inflammatory status)
To assess the correlation between hemoperfusion and positive short-term outcome | 72 hours after finishing the hemoperfusion procedure
  Define as to assess the correlation between hemoperfusion and positive short-term outcome (i.e. an improvement in hemodynamic stability and respiratory status will be combined to report SOFA score)
To assess the correlation between hemoperfusion and positive short-term outcome | 72 hours after finishing the hemoperfusion procedure
  Define as to assess the correlation between hemoperfusion and positive short-term outcome (i.e. an improvement in inflammatory status)
To assess the correlation between hemoperfusion and positive long-term outcome | 28 days
  Define as to assess the correlation between hemoperfusion and positive long-term outcome, defined as patient survival at ICU discharge
The effects of hemoperfusion in combination with other extracorporeal organ support therapies (i.e. ECMO, CRRT) on positive short-term outcome | Immediately after first hemoperfusion procedure in combination with other extracorporeal organ support therapies (i.e. ECMO, CRRT)
  Define as to assess the effects of hemoperfusion in combination with other extracorporeal organ support therapies (i.e. ECMO, CRRT) on positive short-term outcome (i.e. improvement in hemodynamic stability and respiratory status will be combined to report SOFA score)
The effects of hemoperfusion in combination with other extracorporeal organ support therapies (i.e. ECMO, CRRT) on positive short-term outcome | Immediately after first hemoperfusion procedure in combination with other extracorporeal organ support therapies (i.e. ECMO, CRRT)
  Define as to assess the effects of hemoperfusion in combination with other extracorporeal organ support therapies (i.e. ECMO, CRRT) on positive short-term outcome (i.e. improvement in inflammatory status)
The effects of hemoperfusion in combination with other extracorporeal organ support therapies (i.e. ECMO, CRRT) on positive short-term outcome | 72 hours after finishing the procedures with the combination of hemoperfusion and extracorporeal organ support therapy
  Define as to assess the effects of hemoperfusion in combination with other extracorporeal organ support therapies (i.e. ECMO, CRRT) on positive short-term outcome (i.e. an improvement in hemodynamic stability and respiratory status will be combined to report SOFA score)
The effects of hemoperfusion in combination with other extracorporeal organ support therapies (i.e. ECMO, CRRT) on positive short-term outcome | 72 hours after finishing the procedures with the combination of hemoperfusion and extracorporeal organ support therapies (i.e. ECMO, CRRT)
  Define as to assess the effects of hemoperfusion in combination with other extracorporeal organ support therapies (i.e. ECMO, CRRT) on positive short-term outcome (i.e. improvement in inflammatory status)
The effects of hemoperfusion in combination with other extracorporeal organ support therapies (i.e. ECMO, CRRT) on positive long-term outcome | 28 days
  The effects of hemoperfusion in combination with other extracorporeal organ support therapies (i.e. ECMO, CRRT) on positive long-term outcome, defined as patient survival at ICU discharge
To assess the correlation between hemoperfusion and negative short-term outcome | Immediately after first hemoperfusion procedure
  Define as to assess the correlation between hemoperfusion and negative short-term outcome (i.e. initial signs of humoral immune dysregulation (hypogammaglobulinemia defined as a gamma-globulin fraction below 10%) or cascade coagulation disorders (severe thrombocytopenia <15,000 cells/uL or severe bleeding)
To assess the correlation between hemoperfusion and negative short-term outcome | 72 hours after finishing the hemoperfusion procedure
  Define as to assess the correlation between hemoperfusion and negative short-term outcome (i.e. initial signs of humoral immune dysregulation (hypogammaglobulinemia defined as a gamma-globulin fraction below 10%) or cascade coagulation disorders (severe thrombocytopenia <15,000 cells/uL or severe bleeding)
Length of ICU stay | 28 days
  Time spend in the ICU after Seraph 100 therapy session
Length of Hospital stay | 60 days
  Time spend in the hospital after Seraph 100 therapy session
Adverse events | 28 days
  Report of any Seraph 100 therapy related adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Center Zagreb, Zagreb, City of Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No